CLINICAL TRIAL: NCT06108531
Title: Study on the Application of Tumor Exosome Liquid Biopsy in the Early Diagnosis of Pancreatic Cancer
Brief Title: Tumor Exosome Liquid Biopsy Strategy to Diagnose Pancreatic Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yingbin Liu, MD, PhD, FACS, vice-president，Xinhua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China, Shanghai Jiao Tong University School of Medicine
Other Study IDs: IIT-2023-0118
Record Dates: First submitted 2023-10-23; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pancreatic patients: Cases will be the patients with newly-diagnosed pancreatic.
- The controls: Controls will be selected from patients with pancreatitis from the same hospital as the case, matched by gender, race and age (1:1).

INTERVENTIONS:
Other:

SUMMARY:
This is an observational study of patients diagnosed with pancreatic cancer by pathology, with a control group of patients with pathology suggestive of benign pancreatic lesions and normal subjects, and the diagnostic ability of exosomes to identify patients with pancreatic cancer was assessed through the detection of exosomes in the peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of pancreatic cancer confirmed by imaging (case) Diagnosis of chronic pancreatitis confirmed by imaging (hospital control)

Exclusion Criteria:

The pathology diagnosis and imaging does not matched Patients with other malignant tumors Patients with other severe systemic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases will be patients with newly diagnosed pancreatic cancer. Controls will be selected from patients with pancreatitis in the same hospital as the cases, matched by sex, race and age (1:1). A total of 400 patients with gallbladder cancer will be recruited.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of proteins in tumor exosomes from patients with pancreatic cancer | Up to 2 years from start of study
  We will select specific protein A from circulating exosomes of pancreatic cancer patients for further analysis.
The expression of protein A in the circulating exosomes from patients | Up to 2 years from start of study
  By detecting the expression of protein A in circulating exosomes of patients. the ROC curve of A+ circulating exosomes will be compared to clinical standard tumor biomarkers (e.g., CA199) in pancreatic cancer patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Affiliated to Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China